CLINICAL TRIAL: NCT04351815
Title: Short-term Prehabilitation Program : Interest of on Resumption of Function at 2 Months: a Randomized Controlled Study
Brief Title: Short-term Prehabilitation Program : Interest of on Resumption of Function at 2 Months
Acronym: PREHAB-COURT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: As the possible regulatory deadline for the research was exceeded, due to logistical difficulties in setting up the study, and in agreement with the sponsor and the principal investigator, it was decided not to extend the study.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019_0011
Record Dates: First submitted 2020-02-14; First posted 2020-04-17 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Thoracic Diseases; Urologic Diseases
Keywords: prehabilitation
MeSH Terms: conditions — Thoracic Diseases; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short prehabilitation (Experimental): This arm will benefit from a 2 weeks prehabilitation program including a personalized dietetic and physical training program as well as psychological support.
  Interventions: Behavioral: Short term prehabilitation (2 weeks)
- No prehabilitation (Other): This arm will not benefit from a prehabilitation program before surgery. Patients will be told to maintain a regular physical activity without support.
  Interventions: Other: No specific intervention

INTERVENTIONS:
Behavioral: Short term prehabilitation (2 weeks) — * Initial assessment visit with a dietitian, a psychologist, a physiotherapist, a doctor (physical medicine) and a geriatrician (for patients over 75 years old)
  * Patient will be asked to follow a 2 weeks prehabilitation program
  * 2 months post-surgery assessment visit with a dietitian, a psychologist, a physiotherapist, a doctor (physical medicine)
  * 6 months post-surgery assessment visit with a dietitian, a psychologist, a physiotherapist, a doctor (physical medicine)
  Arms: Short prehabilitation
Other: No specific intervention — * Standard care: Initial assessment visit with a dietitian, a psychologist, a physiotherapist, a doctor (physical medicine) and a geriatrician (for patients over 75 years old)
  * Patients will be asked to maintain regular physical activity without support
  * 2 months post-surgery assessment visit with a dietitian, a psychologist, a physiotherapist, a doctor (physical medicine)
  * 6 months post-surgery assessment visit with a dietitian, a psychologist, a physiotherapist, a doctor (physical medicine)
  Arms: No prehabilitation

SUMMARY:
This study aimed to evaluated the interest of a short-term (2 weeks) prehabilitation program compared to no prehabilitation before thoracic or urological surgery

DETAILED DESCRIPTION:
Prehabilitation is a form of global strength training, aims to improve functional capacity before surgery.This preparation compensate for its decrease due to the intervention. This process includes physical training, nutritional and psychological care.

Previous studies consider 4 weeks to be the ideal duration time for such program. However, extended program duration may reduce subject compliance and may not be possible for patient who can not or do not want to postponed their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 55 or over
* Requiring major surgery (thoracic or urological surgery: kidney or bladder) within 15 days after the completion of the inclusion assessment
* Having signed a consent form after a reflection period
* Being affiliated to a Health Insurance plan.

Exclusion Criteria:

* Pregnant, parturient or lactating women
* Persons deprived of their liberty: minors or adults subject to legal protection measures or out of state to express their consent
* Patients (men or women) aged <55 years;
* Inability to walk or initial physical assessment
* Inability to complete questionnaires
* Walk> 450 meters in the 6 minute test
* Patients under guardianship or curators.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Evaluated the change in physical condition of patient following a short prehabilitation compared to the initial assessment (6 minutes walk test) | 7 months
  Change on the 6-minute walk test (distance covered over a time of 6 minutes in meters)
Evaluated the change in physical condition of patient following a short prehabilitation compared to the initial assessment (Borg scale) | 7 months
  Change in the Borg scale (exertion from 0 to 10: 0 meaning no exertion, 10 meaning maximal exertion)

SECONDARY OUTCOMES:
Evaluated the change in cardio-respiratory capacity (VO2 max) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  VO2 Max Testing, measured in milliliters of oxygen used in one minute per kilogram of body weight (milliliter per kilogram per minute).
Evaluated the change in cardio-respiratory capacity (spirometry: maximal voluntary ventilation) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Evolution of Maximal Voluntary Ventilation (MVV in liter per minute).
Evaluated the change in cardio-respiratory capacity (spirometry: vital capacity) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Evolution of Vital Capacity (VC in liter)
Evaluated the change in cardio-respiratory capacity (spirometry: functional residual capacity) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Evolution of Functional residual capacity (FRC in milliliter per kilogram).
Evaluated the change in cardio-respiratory capacity (heart rate) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Heart rate at 40 watt during a cardiac stress test (beats per minute).
Evaluated the change in the muscular mass of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Quadriceps area in square centimeters.
Evaluated the change in the muscular strength of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Hand grip Test (measure in Newton).
Evaluated the change in the body mass (weight) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Weight in kilogram.
Evaluated the change in the body mass (lean mass) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Percentage of lean mass.
Evaluated the change on the psychological state (quality of life) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  SF-36 quality of life scale (eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each items are scored on a 0 to 100 range. A high score defines a more favorable health state).
Evaluated the change on the psychological state (anxiety and depression) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Hospital Anxiety and Depression Scale (HADS)(a fourteen item scale that generates : Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression).
Evaluated the change on the psychological state (fatigue) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Patient-Reported Outcomes Measurement Information System (PROMIS) : PROMIS Fatigue-Short Form (seven items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week on a 5-point Likert scale, ranging from 1 = never to 5 = always).
Evaluated the change on the psychological state (sleep) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Patient-Reported Outcomes Measurement Information System (PROMIS): PROMIS-Sleep Disturbance-Short Form (eight items that measure both the experience problems with sleep and the interference of problems with sleep on daily activities over the past week, ranging from 1 = not at all to 5 = very much).
Evaluated the change on the psychological state (pain) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Patient-Reported Outcomes Measurement Information System (PROMIS): PROMIS Pain Interference - Short Form (six items that measure both the experience of pain and the interference of pain on daily activities over the past week, ranging from 1 = not at all to 5 = very much).
Evaluated the change on the psychological state (geriatric health) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Geriatric health status screening tool (G8 score) (8 questions score between 0 and 17, a higher score indicates a better health status). For geriatric patient only.
Evaluated the change on the psychological state (daily living) of patient following a short prehabilitation at 15 days compared to the initial assessment | 15 days
  Instrumental activities of daily living scale (8 domains of function ranges from 0 (low function, dependent) to 8 (high function, independent))
Evaluate compliance to the prehabilitation program | 15 days
  Overall compliance score regarding physical training, proteins intake, well-being and fatigue (complete, partial or non compliance).
Evaluate post-surgery complications (classification) | 2 months and 6 months
  Classification of complications according to Dindo and Clavien (grades I, II, IIIa, IIIb, IVa, IVb or V).
Evaluate post-surgery complications (length of stay) | 2 months and 6 months
  Length of stay in hospital, in intensive care unit or continuous monitoring unit (number of days).
Evaluate post-surgery complications (mortality) | 2 months and 6 months
  Hospital and 30-day mortality (patient status).
Evaluate post-surgery complications (re-hospitalization) | 2 months and 6 months
  Re-hospitalization in the same hospital within 30 days of discharge from the initial hospitalization (yes/no).
Evaluate post-surgery complications : comparison between predicted complications and actual complications (ARISCAT) | 2 months and 6 months
  ARISCAT score (risk of postoperative respiratory complication considered to be low for a score less than 26, moderate for a score of 26 to 44, and high for a score of 45 or more).
Evaluate post-surgery complications : comparison between predicted complications and actual complications (LEE) | 2 months and 6 months
  LEE score (postoperative cardiac risk (infarction, heart failure, death): 0-1 low risk, 2 significant risk, more than 3 major risk).
Evaluate post-surgery complications : comparison between predicted complications and actual complications (POSPOM) | 2 months and 6 months
  Preoperative Score To Predict Postoperative Mortality (POSPOM) system (scale of 0 to 50 points, with 0 given to patients with the lowest risk).
Evaluate post-surgery complications : comparison between predicted complications and actual complications (Charlson index) | 2 months and 6 months
  Charlson index (22 conditions are assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality. A higher score indicates a higher risk of mortality.)
Evaluate post-surgery complications : comparison between predicted complications and actual complications (POSSUM score) | 2 months and 6 months
  Physiologic and Operative Severity Score for the enUmeration of Mortality and Morbidity score (POSSUM score) (18 factors scored exponentially increasing from 1 to 8. A higher score indicates a higher risk of mortality).
Evaluated the change in cardio-respiratory capacity (6 minutes walk test) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Change on the 6-minute walk test (distance covered over a time of 6 minutes in meters).
Evaluated the change in cardio-respiratory capacity (VO2 max) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  VO2 Max Testing, measured in milliliters of oxygen used in one minute per kilogram of body weight (milliliter per kilogram per minute).
Evaluated the change in cardio-respiratory capacity (spirometry: maximal voluntary ventilation) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Evolution of Maximal Voluntary Ventilation (MVV in liter per minute).
Evaluated the change in cardio-respiratory capacity (spirometry: vital capacity) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Evolution of Vital Capacity (VC in liter).
Evaluated the change in cardio-respiratory capacity (spirometry: functional residual capacity) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Evolution of Functional residual capacity (FRC in milliliter per kilogram).
Evaluated the change in cardio-respiratory capacity (heart rate) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Heart rate at 40 watt during a cardiac stress test (beats per minute).
Evaluated the change in the muscular mass of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Quadriceps area in square centimeters.
Evaluated the change in the muscular strength of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Hand grip Test (measure in Newton).
Evaluated the change in the body mass (weight) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Weight in kilogram.
Evaluated the change in the body mass (lean mass) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Percentage of lean mass.
Evaluated the change on the psychological state (quality of life) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  SF-36 quality of life scale (eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each items are scored on a 0 to 100 range. A high score defines a more favorable health state).
Evaluated the change on the psychological state (anxiety and depression) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Hospital Anxiety and Depression Scale (HADS) (a fourteen item scale that generates : Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression).
Evaluated the change on the psychological state (fatigue) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) : PROMIS Fatigue-Short Form (seven items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week on a 5-point Likert scale, ranging from 1 = never to 5 = always).
Evaluated the change on the psychological state (sleep) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS): PROMIS-Sleep Disturbance-Short Form (eight items that measure both the experience problems with sleep and the interference of problems with sleep on daily activities over the past week, ranging from 1 = not at all to 5 = very much)
Evaluated the change on the psychological state (pain) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS): PROMIS Pain Interference - Short Form (six items that measure both the experience of pain and the interference of pain on daily activities over the past week, ranging from 1 = not at all to 5 = very much).
Evaluated the change on the psychological state (geriatric health) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Geriatric health status screening tool (G8 score) (8 questions score between 0 and 17, a higher score indicates a better health status). For geriatric patient only.
Evaluated the change on the psychological state (daily living) of patient following a short prehabilitation at 2 and 6 months compared to the initial assessment | 2 months and 6 months
  Instrumental activities of daily living scale (8 domains of function ranges from 0 (low function, dependent) to 8 (high function, independent)).
Evaluated the compliance to the prehabilitation program | 2 months and 6 months
  Overall compliance score regarding physical training, proteins intake, well-being and fatigue (complete, partial or non compliance)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch